CLINICAL TRIAL: NCT01434693
Title: A Sequential Dose-Escalation, Double-Blind, Placebo-Controlled, Phase I Study to Evaluate the Safety and Tolerability of Single Doses of 3 Different Doses of Oral CNDO 201 Trichuris Suis Ova Suspension (Tso) in Patients With Crohn's Disease
Brief Title: Safety and Tolerability of Single Doses Oral CNDO 201 Trichuris Suis Ova in Patients With Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coronado Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNDO 201-002
Record Dates: First submitted 2011-09-13; First posted 2011-09-15 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-04

CONDITIONS: Crohn's Disease
Keywords: T. suis ova; Crohn's disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- TSO 500 (Experimental)
  Interventions: Biological: Trichuris suis ova
- TSO 2500 (Experimental)
  Interventions: Biological: Trichuris suis ova
- TSO 7500 (Experimental)
  Interventions: Biological: Trichuris suis ova
- Placebo (Placebo Comparator): single dose
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Trichuris suis ova — single dose
  Arms: TSO 2500; TSO 500; TSO 7500
Other: Placebo
  Arms: Placebo

SUMMARY:
This is a sequential dose-escalation (with up to 3 dose levels of TSO, ie, 500, 2500, and 7500 TSO), randomized (within each of 3 periods, with a ratio of 3:1 for TSO to placebo), double-blind, placebo-controlled study to evaluate the safety of a single dose of oral CNDO-201 Trichuris suis ova suspension, as compared to placebo, in patients with Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 18 to 55 years old.
2. Patient has confirmed diagnosis of Crohn's Disease by established criteria with a minimum disease duration of 3 months.
3. If patient is using concomitant medications, the dose/regimen is stable and remains stable for the two weeks of close observation following TSO administration. Concomitant medications may include: 1) Oral sulfasalazine, mesalazine (5-ASA), or mesalazine derivative, if receiving it for >6 weeks and if receiving the same dose for at least 4 weeks; 2) Oral prednisone up to 15 mg/day, if receiving it for >4 weeks and if receiving the same dose for at least 2 weeks; and 3) Azathioprine or 6-mercaptopurine if receiving it for >3 months and if receiving the same dose for at least 8 weeks.
4. Hemoglobin ≥ 12 g/dL at screening.
5. Normal white blood cell count and normal lymphocyte count at screening.
6. Platelet count > lower limit of normal at screening.
7. For females of childbearing potential, negative serum pregnancy test during the screening period, not breastfeeding for study duration, and willingness to use accepted forms of reliable birth control for study duration [including bilateral tubal ligation, use of oral contraceptives, double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), Depo-Provera®, hormonal implants, partner vasectomy, and total abstinence]. Pregnancy tests are not required (indicate "N/A") for males or females not of childbearing potential (post-menopausal with last menstrual period >1 year ago or total hysterectomy).
8. Patient must have the ability to provide informed consent.

Exclusion Criteria:

1. Patient with ulcerative colitis, indeterminate colitis, or ulcerative proctitis.
2. Bowel surgery in past 6 months.
3. Resection of more than 50 cm of the ileum.
4. Ileostomy colostomy.
5. Septic complications.
6. Patient who is hospitalized or exhibiting signs of toxicity (sepsis), has significant or multiple strictures, or impending obstruction (as evidenced by abdominal distension, severe abdominal tenderness, fever, nausea, vomiting, or tachycardia) or anticipating a need for blood transfusion for gastrointestinal bleeding or in whom surgical intervention may be imminent.
7. Patient with gastrointestinal abscess, perforation, active draining fistulae or fistulae that are considered clinically significant or perianal lesions.
8. Patient with history of colorectal cancer or colorectal dysplasia.
9. Parenteral or tube feeding.
10. Patient with evidence of infectious colitis, e.g., Clostridium difficile, Amoebiasis, Giardia lamblia or stools positive for other enteric pathogens, ova or parasites at Screening.
11. Female patient who is pregnant or breastfeeding or wishing to become pregnant during study participation or unwilling to use birth control.
12. Patient with serum creatinine ≥ 2.0 mg/dL; blood urea nitrogen >40 mg/dL; alkaline phosphatase > 250 U/L; aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 100 U/L; or total bilirubin >1.5 mg/dL.
13. Patient with white blood count <5,000 or >15,000/mm3; platelet count <150,000 per μl; or iron or vitamin B12 deficiency. Correction of lab exclusion is allowed provided that medical condition is not deemed to put patient at risk and stability of result is sustained for a minimum of 30 days.
14. Patient with active hepatitis B virus, hepatitis C virus, liver cirrhosis or portal hypertension, cytomegalovirus, Epstein Barr Virus or herpes simplex virus or is known to be human immunodeficiency virus (HIV) positive.
15. Patient with primary sclerosing cholangitis.
16. Patient with active malignancy or treatment with anticancer drugs in the past 5 years.
17. Patient received cyclosporine, anti-TNF or other immunomodulatory agents other than azathioprine/6-mercaptopurine 12 weeks prior to Screening.
18. Patient received methotrexate 4 weeks prior to Screening.
19. Patient received metronidazole 2 weeks prior to Screening.
20. Patient received non-steroidal anti-inflammatory drugs (NSAIDS) within 2 weeks before Baseline visit for more than 3 consecutive days, except acetylsalicylic acid ≤ 350 mg/d which is allowed.
21. Patient received antibiotic, antifungal or antiparasitic medication in the last 2 weeks prior to Screening and/or would potentially require this during the study treatment period.
22. Patient with history of drug or alcohol abuse within 6 months prior to Screening.
23. Patient with evidence of poor compliance with medical advice and instruction including diet or medication.
24. Patient is unable or unwilling to swallow study medication suspension.
25. Patient with a significant medical condition which puts the patient at risk for study participation and/or for any reason is considered by the Investigator to be an unsuitable candidate to receive CNDO-201 TSO or is potentially put at risk by study procedures.
26. Patients who has participated in another clinical trial within 30 days of Screening for this trial and/or any experimental treatment for this population.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Advanced Clinical Research Institute, Anaheim, California
  - Borland-Groover Clinic, Jacksonville, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Midwest Center for Clinical Research, Lee's Summit, Missouri
  - Center for Digestive & Liver Diseases, Inc, Mexico, Missouri
  - Long Island Clinical Research Associates, LLP, Great Neck, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 clinical sites were initiated, all in the United States, with 6 of these sites enrolling at least one patient. Patients were enrolled from Nov, 2011 to Jan 30, 2012.
Pre-assignment Details: All patients were immediately assigned to a treatment group upon enrollment.
Groups:
- Placebo: Placebo: single dose
- TSO 500; TSO 2500; TSO 7500: Trichuris suis ova : single dose
Period: Overall Study
Arm/Group | Placebo | TSO 500 | TSO 2500 | TSO 7500
Started | 9 | 9 | 9 | 9
Completed | 6 | 9 | 8 | 8
Not Completed | 3 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TSO 500 | TSO 2500 | TSO 7500 | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 9 | 9 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.0 (3.11) | 30.8 (3.19) | 31.1 (3.36) | 36.9 (3.27) | 32.9 (1.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 5 | 18
  Male | 5 | 3 | 6 | 4 | 18
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Comparison of safety and tolerability was performed across the dose levels by evaluating the post-dose tolerability of TSO in patients with Crohn's Disease via incidence of adverse events (i.e. # events) with a specific focus on reported gastrointestinal signs and symptoms
Time Frame: 6 mo
Population: All patients who were randomized were treated according to the protocol and therefore were all included in the Safety Population.
Measure: Number; unit: events
Arm/Group | Placebo | TSO 500 | TSO 2500 | TSO 7500
Number analyzed (Participants) | 9 | 9 | 9 | 9
events | 7 | 4 | 1 | 7

ADVERSE EVENTS:
Arm/Group | Placebo | TSO 500 | TSO 2500 | TSO 7500
Serious Adverse Events (participants affected / at risk) | 2/9 | 0/9 | 0/9 | 1/9
Other Adverse Events (participants affected / at risk) | 5/9 | 4/9 | 1/9 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | TSO 500 (N=9) | TSO 2500 (N=9) | TSO 7500 (N=9)
small intestinal resection (Surgical and medical procedures) | 1 | 0 | 0 | 0 — Patient 01-1011 (Placebo) experienced a small intestinal resection on Day 42 following dosing. This patient discontinued from the study on Day 84 due to symptoms associated with this event.
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Patient 10-2004 (Placebo) experienced abdominal pain with questionable underlying etiology on Day 48.
Crohn's disease flare (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — Patient 09-3011 (TSO 7500) experienced three SAEs: * Crohn's disease flare on Day 85 * Anovaginal fistula on Day 86 * Clostridium difficile infection on Day 86
ANOVULVAR FISTULA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | TSO 500 (N=9) | TSO 2500 (N=9) | TSO 7500 (N=9)
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Vomitting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Mucous stools (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Gastrointestinal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less